CLINICAL TRIAL: NCT04063072
Title: ERAS (Enhanced Recovery After Surgery) Protocol Implementation in Piedmont Region for Hysterectomy of Benign or Malignant Tumors of the Uterus. A Stepped-wedge Cluster Randomized Clinical Trial.
Brief Title: ERAS (Enhanced Recovery After Surgery) Protocol Implementation in Piedmont Region for Hysterectomy.
Acronym: ERAS-Gyneco
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Regina Montis Regalis (Other)
Collaborators: Martini Hospital, Turin, Italy (Other); A.O.U. Città della Salute e della Scienza (Other); Ministry of Health, Italy (Other Government); Regione Piemonte (Other)
Responsible Party: Principal Investigator, Dr. Andrea Puppo, Gynecologists, Ospedale Regina Montis Regalis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ERAS-Gyneco-Piemonte
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Uterine Neoplasms
Keywords: Hysterectomy; Uterine Cervical Neoplasms; Endometrial Neoplasms; Quality Improvement; Perioperative Care; Recovery of Function
MeSH Terms: conditions — Uterine Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Enhanced Recovery After Surgery; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomized clinical trial. Each center starts as control group (usual care) and switch to experimental group (ERAS protocol implementation) according to a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Perioperative care for hysterectomy of benign or malignant tumors of the uterus is managed according to current hospital clinical practice.
- ERAS protocol (Experimental): Perioperative care for hysterectomy of benign or malignant tumors of the uterus is managed according to ERAS protocol.
  Interventions: Procedure: ERAS protocol

INTERVENTIONS:
Procedure: ERAS protocol — In gynecological surgery, the ERAS protocol involves an accurate interview with the patient in the preoperative phase aimed at smoking and alcohol cessation, the reduction of preoperative fasting, the omission of intestinal preparation, the prophylaxis of thromboembolism, a correct antibiotic prophylaxis, the prevention of intraoperative hypothermia, prevention of volume overload, prevention of postoperative nausea and vomiting, very limited use of the nasogastric tube, early removal of the urinary catheter, multimodal analgesia to minimize opiate consumption, early postoperative mobilization and early post-operative feeding, to promote rapid recovery of gastro-intestinal functions.
  Other Names: ERAS (Enhanced Recovery After Surgery) protocol
  Arms: ERAS protocol

SUMMARY:
The study assesses the impact on quality of care of implementing the ERAS (Enhanced Recovery After Surgery) protocol for hysterectomy of benign or malignant tumors of the uterus in the network of public hospitals in the Regione Piemonte (North-West Italy). Every hospital is a cluster entering the study treating patients according to its current clinical practice. On the basis of a randomized order, each hospital switches from current clinical practice to the adoption of the ERAS protocol.

DETAILED DESCRIPTION:
ERAS (Enhanced Recovery After Surgery) protocol is a multimodal perioperative care pathways designed to achieve early recovery after surgical procedures by maintaining preoperative organ function and reducing the profound stress response following surgery. Even if efficacy and safety of ERAS protocol in gynaecological surgery is well-established in the literature, its implementation is limited to few selected centres in Piemonte. The aim of the study is to extend the implementation of the ERAS protocol to whole regional network of hospitals. Specific objectives are to estimate its impact on different dimensions of quality of care, including length of stay, complications and patient satisfaction, and to identify possible barriers or facilitating factors.

ELIGIBILITY:
Inclusion Criteria:

* All the hospital wards within the Piemonte Region performing hysterectomy.
* All the patients receiving an elective hysterectomy for benign or malignant tumors of the uterus.

Exclusion Criteria:

* Hospital wards performing less than 20 expected cases per year
* Emergency hysterectomy
* Hysterectomy for pelvic floor disorders
* High severity cases not allowing ERAS protocol implementation (i.e. American Society of Anesthesiologists score: ASA V).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecological surgery
Enrollment: 1800 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay | 12 days after admission
  Mean length of stay calculated as difference between date of discharge and date of admission of the hospitalization for surgery, excluding length of stay >12 days (98th percentile of the expected distribution).

SECONDARY OUTCOMES:
Length of stay >12 days | 30 days after admission
  Rate of patients with a length of stay >12 days
Recovery after surgery | 24 hours after surgery
  Score of quality of recovery at 24 hours after surgery, assessed with the questionnaire Quality of Recovery (QoR-15), a 15-items instrument, with responses recorded on a 11-point Likert-type scale form 0 (worst scenario) to 10 (best scenario) and an overall score ranging from 0 (poor recovery) to 150 (excellent recovery).
  A visual analogue scale (VAS), ranging from 0 (worst imaginable health state) to 10 (worst imaginable health state) is also supplied as summary evaluation.
Complications | 30 days after discharge
  Rate of surgical and medical complication after surgery For surgical complications: Comprehensive Complication Index
Transfer to intensive care unit | 30 days after surgery
  Rate of transfers to intensive care unit after surgery
Emergency visits after discharge | 30 days after discharge
  Rate of emergency visit in the first month after discharge
Hospital admissions after discharge | 30 days after discharge
  Rate of new admissions in the first month after discharge
Reintervention | 30 days after surgery
  Rate of reintervention in the first month after surgery, excluding planned interventions
Patients' satisfaction | 15 days after discharge
  Score of patients' satisfaction measured 2 weeks after discharge, assessed with the questionnaire Surgical Satisfaction Questionnaire (SSQ8) supplied by telephone. SSQ8 is a 8-items instrument, with responses recorded on a 5-point Likert-type scale from 0 (worst scenario) to 4 (best scenario) and an overall score ranging from 0 (very unsatisfied) to 32 (very satisfied).
Healthcare costs | 30 days after discharge
  Mean healthcare costs from pre admission visit to 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Giovannino Ciccone, MD, Study Chair — Azienda Ospedaliera Universitaria Città della Salute e della Scienza di Torino
Locations (1):
- Ospedale Regina Montis Regalis, Mondovì, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Derived] Piovano E, Puppo A, Camanni M, Castiglione A, Delpiano EM, Giacometti L, Rolfo M, Rizzo A, Zola P, Ciccone G, Pagano E; ERAS-Gyneco Piemonte Group. Implementing Enhanced Recovery After Surgery for hysterectomy in a hospital network with audit and feedback: A stepped-wedge cluster randomised trial. BJOG. 2024 Aug;131(9):1207-1217. doi: 10.1111/1471-0528.17797. Epub 2024 Feb 25. PMID 38404145
- [Derived] Piovano E, Pagano E, Del Piano E, Rinaldi F, Palazzo V, Coata P, Bongiovanni D, Rolfo M, Ceretto Giannone L, Veliaj D, Camanni M, Puppo A, Ciccone G; ERAS-Gyneco Piemonte group. Implementation of the ERAS (Enhanced Recovery After Surgery) protocol for hysterectomy in the Piedmont Region with an audit&feedback approach: Study protocol for a stepped wedge cluster randomized controlled trial. A study of the EASY-NET project. PLoS One. 2022 May 27;17(5):e0268655. doi: 10.1371/journal.pone.0268655. eCollection 2022. PMID 35622826
- [Derived] Chau JPC, Liu X, Lo SHS, Chien WT, Hui SK, Choi KC, Zhao J. Perioperative enhanced recovery programmes for women with gynaecological cancers. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD008239. doi: 10.1002/14651858.CD008239.pub5. PMID 35289396